CLINICAL TRIAL: NCT00862823
Title: The Stability and Bioequivalence of Tenofovir, Emtricitabine and Efavirenz (Atripla) in an Extemporaneously Prepared Oral Liquid Formulation Compared With the Commercially Available Tablet Formulation
Brief Title: The Bioequivalence of Atripla in an Oral Liquid Formulation Compared With the Tablet Formulation in Healthy Volunteers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Principal Investigator, Jennifer King, Principal Investigator, University of Alabama at Birmingham
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: F081030003
Record Dates: First submitted 2009-03-13; First posted 2009-03-17 (Estimated); Results first posted 2012-09-14 (Estimated); Last update posted 2012-09-14 (Estimated); Status verified 2012-06

CONDITIONS: Healthy
Keywords: Healthy Volunteers
MeSH Terms: interventions — Tenofovir; Emtricitabine; efavirenz; Tablets

ARMS (2):
- Atripla Tablet (Active Comparator): Drug exposure after administration of Atripla Tablet
  Interventions: Drug: tenofovir, emtricitabine and efavirenz fixed dose tablet
- Atripla Liquid (Experimental): Drug exposure after administration of an extemporaneously prepared liquid formulation of Atripla
  Interventions: Drug: tenofovir, emtricitabine and efavirenz tablet added to solution

INTERVENTIONS:
Drug: tenofovir, emtricitabine and efavirenz fixed dose tablet — Atripla contains 300mg of tenofovir, 200mg of emtricitabine and 600mg of efavirenz
  Arms: Atripla Tablet
Drug: tenofovir, emtricitabine and efavirenz tablet added to solution — Atripla contains 300mg of tenofovir, 200mg of emtricitabine and 600mg of efavirenz
  Arms: Atripla Liquid

SUMMARY:
The primary objective of this study is to determine the average bioequivalence of tenofovir, emtricitabine and efavirenz in an extemporaneously prepared oral liquid formulation (test formulation) compared with the commercially available tablet formulation (reference formulation). The study is designed as an open-label, randomized, 2-period, 2-treatment, 2-sequence, single-dose intensive pharmacokinetic study conducted in healthy volunteers. Subjects will be randomized to receive the Atripla tablet (reference formulation) or the Atripla tablet crushed and mixed in OraSweet solution (test formulation) on Study Day 1. Subjects will undergo a 12-hour intensive pharmacokinetic evaluation after ingesting a single dose of either the test or reference formulation. On days 2 and 3, subjects will provide an additional pharmacokinetic sample 24 and 48 hours post dose, respectively. Subjects will complete a washout period from day 2 to day 14 during which no study drugs will be ingested. On day 14, subjects will ingest either the reference or test formulation (opposite of the formulation received on Study Day 1). All subjects will undergo another 12-hour intensive pharmacokinetic evaluation. On days 16 and 17 subjects will provide an additional pharmacokinetic sample 24 and 48 hours post dose, respectively. Adverse events and concomitant medications will be documented throughout the study.

The sample size is 16 and is based upon a 10% drop-out rate (i.e. due to lost to follow-up, treatment discontinuation, etc.). Since the investigators are expecting two subjects not to complete the study, the investigators expect 14 evaluable subjects. If the discontinuation rate is greater than 10%, the investigators will continue to enroll until the investigators get 14 evaluable subjects. The primary endpoint is to determine average bioequivalence for test and reference formulations of tenofovir, emtricitabine and efavirenz according to the FDA guidance on bioequivalence testing. The ratio of the test to reference formulation mean Cmax and AUC24 for each drug and the 90% confidence interval around each mean ratio will be determined. Average bioequivalence will be met if 90% confidence intervals around the Cmax, and AUC24 mean ratios for each drug falls within the FDA's predefined limits of 0.80 to 1.25.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥19 and ≤65, HIV-1 negative, Able to give consent, Non-smoking,Screening EKG within normal limits, Females of childbearing potential must have a negative pregnancy test at screening and agree to use a double-barrier method of contraception throughout the study period.

Exclusion Criteria:

* Subjects receiving any prescription or over-the-counter products will be excluded from the study. Subjects using any form of recreational drugs will be excluded. Subjects who have any of the following laboratory abnormalities within 30 days of study entry will be excluded:

  * SGOT (AST)/SGPT (ALT) > 3 x upper limits of normal (ULN) (Subjects with liver disease are allowed to enroll unless their AST/ALT levels are greater than three times ULN)
  * Bilirubin > 2.5 x ULN
  * Amylase > 2 x ULN
  * Absolute Neutrophil Count < 1000 x 103/L
  * Hgb < 9.0 g/dl
  * Platelets <50,000 cells/mm3
  * Serum Creatinine > 2.5 mg/dl

Ages: 19 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2009-02; Primary Completion 2010-02 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer R King, PharmD, Principal Investigator — University of Alabama at Birmingham
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States

REFERENCES:
- [Result] King J, McCall M, Cannella A, Markiewicz MA, James A, Hood CB, Acosta EP. A randomized crossover study to determine relative bioequivalence of tenofovir, emtricitabine, and efavirenz (Atripla) fixed-dose combination tablet compared with a compounded oral liquid formulation derived from the tablet. J Acquir Immune Defic Syndr. 2011 Apr 15;56(5):e130-2. doi: 10.1097/qai.0b013e31820eefbe. No abstract available. PMID 22046602

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Healthy volunteers recruited in Birmingham, AL from March 2009 and August 2009
Groups:
- Tablet First, Then Liquid: Single dose of Atripla tablet in first intervention period and Single dose of Atripla liquid in second intervnetion period
- Liquid First, Then Tablet: Single dose of Atripla liquid in first intervention period and single dose of Atripla tablet in second intervnetion period
Period: First Intervention
Arm/Group | Tablet First, Then Liquid | Liquid First, Then Tablet
Started | 6 | 10
Completed | 5 | 9
Not Completed | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1
Period: Washout Period of 2 Weeks
Arm/Group | Tablet First, Then Liquid | Liquid First, Then Tablet
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Tablet First, Then Liquid | Liquid First, Then Tablet
Started | 5 | 9
Completed | 5 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Entire Study Population: Includes groups randomized to receive tablet first and liquid first
Arm/Group | Entire Study Population
Number analyzed (Participants) | 16
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 16
  >=65 years | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 33.3 (10.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 9
Region of Enrollment [Number; unit: participants]
  United States | 16

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration Time Curve for Tenofovir, Emtricitabine and Efavirenz
Description: The area under the concentration time curve for tenofovir, emtricitabine and efavirenz
Time Frame: 17 days
Population: US Food and Drug Administration. Guidance for Industry: Bioavailability and Bioequivalence Studies for Orally Administered Drug ProductsdGeneral Considerations. Rockville, MD: United States Food and Drug Administration Center for Drug Evaluation and Research.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg*hr/mL
Groups:
- Atripla Tablet; Atripla Liquid: Includes groups randomized to receive tablet first and liquid first
Arm/Group | Atripla Tablet | Atripla Liquid
Number analyzed (Participants) | 14 | 14
mg*hr/mL
  Efavirenz AUC | 58.7 (57.5) | 56.7 (80)
  Emtricitabine AUC | 10.9 (24.7) | 10.8 (15.9)
  Tenofovir AUC | 1.8 (29.2) | 2.2 (36.3)
Statistical Analysis 1: Comparison: Atripla Tablet vs Atripla Liquid; Test type: Non-Inferiority or Equivalence — The sample size was determined so there was an 80% chance that a 90% pairwise interval for 2 equivalent formulations would satifsy the FDA criteria for AUC and Cmax of log (0.8), log (1.2); p < 0.05, log transformation — Bioequivalent measurew were log-transformed; Geometric Mean Ratio = 0.97

2. Primary Outcome: Maximum Concentration for Tenofovir, Emtricitabine and Efavirenz
Description: The maximum concentration for tenofovir, emtricitabine and efavirenz
Time Frame: 17 days
Population: as for outcome 1
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: mg/L
Arm/Group | Atripla Tablet | Atripla Liquid
Number analyzed (Participants) | 14 | 14
mg/L
  Efavirenz Cmax | 1.5 (39) | 1.3 (28.8)
  Emtricitabine Cmax | 1.8 (32.3) | 2.1 (21)
  Tenofovir Cmax | 0.3 (27.7) | 0.2 (47.8)

ADVERSE EVENTS:
Arm/Group | Entire Study Population
Serious Adverse Events (participants affected / at risk) | 0/16
Other Adverse Events (participants affected / at risk) | 0/16

LIMITATIONS AND CAVEATS:
Efavirenz exposure was highly variable and relative bioequivalence for efavirenz may have been more appropriately assessed with a larger sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No